CLINICAL TRIAL: NCT02642276
Title: Influence of Different Types of Exercise Training on Selected Cardiovascular Parameters in Individuals With Peripheral Arterial Disease
Brief Title: Exercise Training in Individuals With Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Borut Jug, Assistant Professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKCLRehab0022015
Record Dates: First submitted 2015-12-20; First posted 2015-12-30 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: exercise training
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Exercise

ARMS (3):
- Maximal walking group (Active Comparator): Patients to be randomized to the 'maximal walking group' will have exercise training sessions 3 times per week for a period of 12 weeks. They will undergo an exercise training programme consisting of 60 minutes of repetitive interval muscle training/walking up to the point of pain-free walking distance.
  Interventions: Other: Exercise training
- Submaximal walking group (Active Comparator): Patients to be randomized to the 'submaximal walking group' will have exercise training sessions 3 times per week for a period of 12 weeks. They will undergo an exercise training programme consisting of 60 minutes of repetitive interval muscle training/walking up to 2/3 of pain-free walking distance.
  Interventions: Other: Exercise training
- Usual care group (No Intervention): Patients to be randomized to the 'usual care group' will undergo standard care for 12 weeks.

INTERVENTIONS:
Other: Exercise training — Patients to be randomized to the 'maximal walking group' or 'submaximal group' will undergo exercise training sessions 3 times per week for a period of 12 weeks.
  Arms: Maximal walking group; Submaximal walking group

SUMMARY:
In this controlled trial, patients with peripheral arterial disease will be randomized to either maximal walking, submaximal walking, or usual care groups.

DETAILED DESCRIPTION:
Exercise training (walking) is a recommended therapeutic intervention for patients with peripheral arterial disease (PAD). Studies have shown that exercise training improves walking distance, pain-free walking distance, endothelial function and quality of life in these patients. However, to date the most effective exercise training option in terms of improvement of cardiovascular parameters has not been clearly identified. In this controlled trial, patients with PAD will be randomized to either maximal walking group, submaximal walking group, or usual care. The aim of the study is to compare the effect of maximal vs. submaximal walking training programmes on i) walking ability, ii) vascular function, iii) arrhythmogenic potential, iv) parameters of inflammation, hemostasis and heart failure severity, v) health-related quality of life in individuals with PAD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed peripheral arterial disease,
* Fontaine stage II,
* not included in a cardiovascular rehabilitation programme for at least 3 months.

Exclusion Criteria:

* contraindications for physical activity,
* uncontrolled dysrhythmias,
* uncontrolled heart failure (New York Heart Association (NYHA) stage IV),
* unstable coronary or other arterial disease,
* intellectual development disorder,
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change of maximum walking distance, measured in metres | 3 months
  Determined by treadmill walking test.

SECONDARY OUTCOMES:
Change of flow-mediated dilatation of the brachial artery, measured in % | 3 months
Change of the arterial stiffness coefficient | 3 months
Change of the value of blood C-reactive protein, measured in mg/l | 3 months
Change of the value of blood fibrinogen, measured in g/l | 3 months
Change of the value of blood D-dimer, measured in microg/l | 3 months
Change of the value of blood N terminal-proBNP, measured in ng/l | 3 months
Change of from-the-questionnaire-obtained quality of life, measured in points | 3 months
Change of the ECG waves | 3 months
  Estimated with digital high-resolution ECG
Change of the heart rate variability | 3 months
  Estimated with digital high-resolution ECG

CONTACTS AND LOCATIONS:
Overall Officials: Borut Jug, MD, Ph.D., Principal Investigator — University Medical Centre Ljubljana, Slovenia
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Januszek R, Mika P, Konik A, Petriczek T, Nowobilski R, Nizankowski R. Effect of treadmill training on endothelial function and walking abilities in patients with peripheral arterial disease. J Cardiol. 2014 Aug;64(2):145-51. doi: 10.1016/j.jjcc.2013.12.002. Epub 2014 Jan 14. PMID 24438856
- [Background] Mika P, Konik A, Januszek R, Petriczek T, Mika A, Nowobilski R, Nizankowski R, Szczeklik A. Comparison of two treadmill training programs on walking ability and endothelial function in intermittent claudication. Int J Cardiol. 2013 Sep 30;168(2):838-42. doi: 10.1016/j.ijcard.2012.10.003. Epub 2012 Oct 30. PMID 23117015
- [Background] Delaney CL, Miller MD, Allan RB, Spark JI. The impact of different supervised exercise regimens on endothelial function in patients with intermittent claudication. Vascular. 2015 Dec;23(6):561-9. doi: 10.1177/1708538114558329. Epub 2014 Nov 18. PMID 25406267
- [Background] McDermott MM, Greenland P, Green D, Guralnik JM, Criqui MH, Liu K, Chan C, Pearce WH, Taylor L, Ridker PM, Schneider JR, Martin G, Rifai N, Quann M, Fornage M. D-dimer, inflammatory markers, and lower extremity functioning in patients with and without peripheral arterial disease. Circulation. 2003 Jul 1;107(25):3191-8. doi: 10.1161/01.CIR.0000074227.53616.CC. Epub 2003 Jun 16. PMID 12810614
- [Background] Mika P, Wilk B, Mika A, Marchewka A, Nizankowski R. The effect of pain-free treadmill training on fibrinogen, haematocrit, and lipid profile in patients with claudication. Eur J Cardiovasc Prev Rehabil. 2011 Oct;18(5):754-60. doi: 10.1177/1741826710389421. Epub 2011 Feb 9. PMID 21450630
- [Background] Schlager O, Hammer A, Giurgea A, Schuhfried O, Fialka-Moser V, Gschwandtner M, Koppensteiner R, Steiner S. Impact of exercise training on inflammation and platelet activation in patients with intermittent claudication. Swiss Med Wkly. 2012 Aug 14;142:w13623. doi: 10.4414/smw.2012.13623. eCollection 2012. PMID 22893497
- [Background] Parmenter BJ, Dieberg G, Phipps G, Smart NA. Exercise training for health-related quality of life in peripheral artery disease: a systematic review and meta-analysis. Vasc Med. 2015 Feb;20(1):30-40. doi: 10.1177/1358863X14559092. Epub 2014 Nov 28. PMID 25432991
- [Background] Gardner AW, Montgomery PS, Flinn WR, Katzel LI. The effect of exercise intensity on the response to exercise rehabilitation in patients with intermittent claudication. J Vasc Surg. 2005 Oct;42(4):702-9. doi: 10.1016/j.jvs.2005.05.049. PMID 16242558
- [Derived] Novakovic M, Krevel B, Rajkovic U, Vizintin Cuderman T, Jansa Trontelj K, Fras Z, Jug B. Moderate-pain versus pain-free exercise, walking capacity, and cardiovascular health in patients with peripheral artery disease. J Vasc Surg. 2019 Jul;70(1):148-156. doi: 10.1016/j.jvs.2018.10.109. Epub 2019 Mar 25. PMID 30922760